CLINICAL TRIAL: NCT02961452
Title: Phenotypical Characterization of Peanut Allergic Children With Differences in Cross-allergy to Tree Nuts and Other Legumes
Brief Title: Phenotypical Characterization of Peanut Allergic Children
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-066
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Nut Hypersensitivity; Child; Legumes Allergy; Tree Nut Allergy; Allergy Cross Reaction
MeSH Terms: conditions — Nut Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peanut allergic children
  Interventions: Other: Cross reaction detection

INTERVENTIONS:
Other: Cross reaction detection

SUMMARY:
Peanut allergy (PA) has been well studied and its prevalence was estimated up to 1.3% in Europe. Tree nut (TN) allergy and PA are clinically similar and often coexist, TN allergy prevalence ranged from 0.05 to 4.9 %. TN allergy is longlasting and nearly all TN have been associated with fatal allergic reactions . Other legumes or TN also contain seed storage protein orthologs of the globulins (Ara h1, Ara h 3) and 2S albumins (Ara h 2) of peanut, susceptible to provoke allergic reactions, but cross-reactivity to TN and other legumes in PA patients could also appear through primarily sensitization. These possible IgE-binding cross-reactions bring to recommend the avoidance of TN and other legumes which have never been eaten in PA children. In this context, diagnosis work-up of relevant cross-allergy versus asymptomatic cross-sensitization will impact directly children's health-related quality of life (HRQL).

When physicians suspect food allergy, many parameters have to be considered, such as clinical background, clinical history, type of symptoms related to the suspected food and cross-allergy to other foods. Then, to objectively confirm a food allergy and to assess its severity (related to the threshold reactive dose and symptoms), an oral food challenge (OFC) is demanded, and double-blind placebo-controlled food challenge (DBPCFC) is considered as "the gold standard".

Although OFC are more and more available in the diagnosis of PA, the assessment of cross-allergy to every single allergenic TN and legumes requires full allergy work-up and often many years of follow-up. Few studies investigated cross-allergy to TN and other legume, with rates of cross-allergy to TN between 28% and 50%. However, targeting patients with severe or cross-allergic phenotypes would greatly assist the allergist in management and follow-up of PA patients (i.e., planning OFC to cross-reactive food).

Our main objective is to identify different disease phenotypes of PA children with cluster analysis. This statistical approach has never been performed to identify cross-allergic phenotypes. We also will describe cross-allergy in PA and will identify possible risk factors for cross-allergy to TN and other legumes in PA children.

ELIGIBILITY:
Inclusion Criteria:

* Child evaluated at the allergy Unit of Saint Vincent Hospital of Lille (France) from March 2004 to May 2016
* Peanut allergy proven with a double-blind placebo-controlled food challenge

Exclusion Criteria:

* Patients who had incomplete evaluation for major peanut component at the time of their double-blind placebo-controlled food challenge to peanut.
* All patients refusing Oral Food Challenge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with peanut allergy who had a complete evaluation about cross-allergy to Tree Nuts and other legumes
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Double-blind placebo-controlled food challenge Test for determination of type of allergic reaction | at inclusion
  After the test (DBPCFC) the type of allergic reaction will be registered: asthma and allergic rhinitis (AR)
Double-blind placebo-controlled food challenge Test for determination of threshold reactive dose | at inclusion
Measure of specific IgEs for the peanut component Ara h 1, Ara h 2, Ara h 3 | at inclusion
Oral food challenge test for diagnosis of tree nuts and/or other legumes allergies | through the study completion

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Cousin, MD, Principal Investigator — GHICL

IPD SHARING:
Plan to Share IPD: No